CLINICAL TRIAL: NCT02107573
Title: Will Routine Suprascapular Nerve Release During Arthroscopic Rotator Cuff Repair Improve Patient Outcomes?
Brief Title: Comparing the Outcomes Between Rotator Cuff Repair With and Without Suprascapular Nerve Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB13-0099
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Tear
Keywords: Randomized Controlled Trial; Rotator Cuff Tear; Suprascapular Nerve; Decompression; Shoulder Surgery
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotator cuff repair without Suprascapular Nerve decompression (Active Comparator): approximately 17 subjects in the study will receive traditional rotator cuff repair surgical intervention with no suprascapular nerve decompression surgical intervention
  Interventions: Procedure: Rotator Cuff Repair without Suprascapular Nerve decompression
- Rotator Cuff Repair with Suprascapular Nerve decompression (Active Comparator): approximately 17 subjects in the study will undergo rotator cuff repair with arthroscopic suprascapular nerve decompression surgical intervention
  Interventions: Procedure: Rotator Cuff Repair with Suprascapular Nerve decompression

INTERVENTIONS:
Procedure: Rotator Cuff Repair without Suprascapular Nerve decompression — Traditional rotator cuff repair without Suprascapular nerve decompression
  Arms: Rotator cuff repair without Suprascapular Nerve decompression
Procedure: Rotator Cuff Repair with Suprascapular Nerve decompression — Traditional rotator cuff repair with Suprascapular nerve decompression
  Arms: Rotator Cuff Repair with Suprascapular Nerve decompression

SUMMARY:
The purpose of the study is to compare the differences in outcome between the traditional rotator cuff repair surgery and rotator cuff repair with suprascapular nerve decompression surgery.

DETAILED DESCRIPTION:
The suprascapular nerve is intimately related to the function and likely recovery of the rotator cuff musculature. Retracted rotator cuff tears have recently been shown to effect both the physical path in which the suprascapular nerve travels, as well as its physiologic function.

This study will be a randomized control trial with long term follow up that will add to and elaborate on the positive outcomes reported in other trials. Patients that have a rotator cuff tears with greater than or equal to 1 cm of retraction that have failed conservative treatment and require operative repair will qualify for the study. They will be randomized into two arms: In one arm, patients will undergo suprascapular nerve release immediately after their rotator cuff repair; they will be compared to patients that have rotator cuff repair with no release of the nerve. Post operatively, at different time intervals, patients will be expected to fill out multiple standardized, well established surveys that assess the patients pain level and shoulder function.

ELIGIBILITY:
Inclusion Criteria:

* Reparable full thickness supraspinatus and or infraspinatus rotator cuff tears regardless of retraction

Exclusion Criteria:

* Patients less than 18 years of age
* Irreparable rotator cuff tears

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | one year
  The scale measures pain from 0 to 10 and also includes a questionnaire for assessing the activity of daily living.

SECONDARY OUTCOMES:
Constant Shoulder Score | one year
  It includes pain score, functional assessment, range of motion and strength measures

CONTACTS AND LOCATIONS:
Overall Officials: Lewis L Shi, MD, Principal Investigator — University of Chicago; Jason Koh, MD, Principal Investigator — Northshore University
Locations (2):
- United States (2):
  - The University of Chicago Medical Center, Chicago, Illinois
  - Northshore University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No